CLINICAL TRIAL: NCT07130383
Title: An Open-label Phase II Clinical Study of MHB036C for Injection Combined With MHB039A for Injection in Patients With Advanced Breast Cancer or Other Advanced Malignant Solid Tumors
Brief Title: A Study of MHB036C Combined With MHB039A in Patients With Advanced Breast Cancer or Other Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MHB036C-E-202
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Advanced Breast Cancer; Advanced Malignant Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Safety run-in phase: cohort 1 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Safety run-in phase: cohort 2 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose expansion phase: cohort 1 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose expansion phase: cohort 2 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose expansion phase: cohort 3 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose expansion phase: cohort 4 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose expansion phase: cohort 5 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration.
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection

INTERVENTIONS:
Drug: MHB036C for Injection — Intravenous administration
Drug: MHB039A for Injection — Intravenous administration

SUMMARY:
This is an open-label, multicenter Phase II study of MHB036C combined with MHB039A in patients with advanced Breast Cancer or other advanced malignant solid tumors. The study was designed to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of MHB036C and MHB039A combination therapy.

DETAILED DESCRIPTION:
This phase II clinical trial of MHB036C and MHB039A combination therapy comprises two parts: a safety run-in phase and an indication expansion phase. The safety run-in phase includes a dose escalation part and an optional PK expansion part. The primary objectives are to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of MHB036C combined with MHB039A in patients with advanced solid tumors. The optional PK expansion part is allowed to enroll additional patients at any non-DLT dose levels that have completed DLT (dose-limiting toxicity) evaluation.

Based on the safety, PK, and preliminary efficacy data from the safety run-in phase, the sponsor will initiate the indication expansion phase at selected dose levels. This phase is an open-label, multicenter, multi-cohort study designed to further evaluate the efficacy and safety of MHB036C and MHB039A combination therapy in patients with advanced breast cancer and other specific types of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agrees to participate in the study and signs the informed consent form.
2. Age ≥ 18 and ≤75 years, no restriction on gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Estimated life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed locally advanced or metastatic advanced solid tumors.
6. At least one measurable lesion per RECIST v1.1 criteria.
7. Adequate bone marrow reserve and organ function.
8. Eligible participants of childbearing potential (males and females) must agree to take highly reliable contraceptive measures with their partners during the study and within at least 12 weeks after the last dose.

   -

Exclusion Criteria:

1. History of ≥2 primary malignancies within 5 years prior to informed consent.
2. Received anti-tumor treatment within 4 weeks or within the 5 half-lives of the previous treatment (whichever is shorter) before dosing.
3. Medication of other unmarketed investigational drugs or therapies within 4 weeks before dosing.
4. Undergone major organ surgery (excluding biopsy) or significant trauma within 4 weeks before dosing or requiring elective surgery during the study.
5. Vaccinated with attenuated live vaccines within 4 weeks before dosing.
6. Treated with with systemic corticosteroids within 14 days before dosing.
7. Central nervous system metastasis.
8. Uncontrolled third-space effusion.
9. Serious cardiovascular or cerebrovascular diseases.
10. Severe lung disease affecting pulmonary function.
11. Active infection requiring systemic therapy.
12. Known hypersensitivity or delayed allergic reaction to the investigational product or its components.
13. Drug abuse or other medical/psychiatric condition that may interfere with study participation or results.
14. Known alcohol or drug dependence.
15. Pregnant or breastfeeding women, or individuals planning to conceive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
(Dose-Expansion Stage): Objective tumor response (ORR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).

SECONDARY OUTCOMES:
Duration of response (DOR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Disease control rate (DCR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose].
Progression-free survival (PFS) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). PFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to PD or death from any cause.
Overall survival (OS) | Baseline up until death up to approximately 5 years
  OS was defined as the time from random assignment or first dose to death from any cause.
Incidence and severity of adverse events (AEs) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years.
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0].
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | From pre-dose to 22 days after the first dose
  The PK parameters at different time points include:Area Under the Concentration-Time Curve (AUC).
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | From pre-dose to 22 days after the first dose
  The PK parameters at different time points include:Maximum Plasma Concentration (Cmax).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No